CLINICAL TRIAL: NCT00205218
Title: Validation of Methods to Estimate Body Fat
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-1998-0373
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2007-04

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate various methods for estimating body composition in human subjects. Each subject is evaluated by several methods that are then compared to a criterion value. We hypothesize that the prediction method will yield the same result as the criterion value. The risks to subjects are minimal and all techniques are routinely performed.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female (pre-menopausal) volunteers

Exclusion Criteria:

* post-menopausal and pregnant women

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1998-11; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Clark, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States